CLINICAL TRIAL: NCT06712836
Title: A Phase 2b, Multi-Center, Randomized, Placebo-Controlled Double-Blind Study to Investigate the Safety and Efficacy of Once-Weekly MET097 in Participants With Obesity and Overweight (VESPER-1)
Brief Title: A Phase 2b Study to Examine the Safety and Efficacy of Once-Weekly MET097 in Adults With Obesity or Overweight
Acronym: VESPER-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Metsera, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MET097-24-201
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-10

CONDITIONS: Obesity; Overweight or Obesity
Keywords: Overweight; GLP-1
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MET097 Active (Experimental): MET097 will be administered at four different dose levels subcutaneously once-weekly without titration. The extension phase includes dosing regimens that are less frequent than weekly.
  Interventions: Drug: MET097
- Placebo (Placebo Comparator): Sterile 0.9% (w/v) saline will be used as placebo treatment during the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MET097 — MET097 is an ultra-long-acting, fully-biased analog of human GLP-1.
  Arms: MET097 Active
Drug: Placebo — Sterile 0.9% (w/v) saline will be used as placebo treatment during the study.
  Arms: Placebo

SUMMARY:
This study is designed to test how well MET097, an active drug, works to treat individuals with obesity or overweight when compared to placebo. MET097 or placebo will be given to individuals weekly for 28 weeks. If an individual is assigned to MET097 they will receive one of four different dose levels. Participants who have completed the first 28 weeks may participate in an exploratory extension study.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled study to investigate the efficacy and safety of four different dose levels of MET097 vs. placebo for body weight loss in adult participants with obesity or overweight (body mass index [BMI] 27 to 50 kg/m2, aged 18 to 70), after 28 weeks with once weekly dosing. Participants who have completed the first 28 weeks may participate in an exploratory extension study that includes less frequent dosing regimens. After the dosing period, there is an additional post-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) at Screening of:

  * BMI ≥30 kg/m2 and ≤50.0 kg/m2 (can have the weight-related co-morbidities listed below)
  * BMI ≥27.0 kg/m2 to <30.0 kg/m2 with at least one of the following weight-related co-morbidities:

    1. Hypertension: on blood pressure (BP)-lowering medication or having systolic BP ≥130 mmHg or diastolic BP ≥80 mmHg at Screening
    2. Dyslipidemia: on lipid-lowering medication or having low-density lipoprotein cholesterol (LDL-C) ≥160 mg/dL (4.1 mmol/L) or triglycerides ≥150 mg/dL (1.7 mmol/L), or high-density lipoprotein-cholesterol (HDL-C) <40 mg/dL (1.0 mmol/L) for men or HDL-C <50 mg/dL (1.3 mmol/L) for women at Screening

Stable body weight (increase or decrease ≤5 kg) within 3 months prior to Screening

Exclusion Criteria:

* Diagnosis of diabetes (T1DM or T2DM) or glycated hemoglobin A1c (HbA1c) ≥ 6.5% or fasting plasma glucose >125 mg/dL.
* Estimated glomerular filtration rate (eGFR) <75 mL/min/1.73 m2
* History of pancreatitis
* Family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* History of significant active or unstable major depressive disorder (MDD) or other severe psychiatric disorder within the last 2 years
* Any lifetime history of a suicide attempt.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in body weight at Week 28 | Baseline (Week 0) through Week 28 (Day 197)
  Evaluate the efficacy of once-weekly MET097 on body weight after 28 once-weekly doses compared to placebo.

SECONDARY OUTCOMES:
Weight reduction (weight loss) from baseline that is ≥ 5% | Baseline (Week 0) through Week 28 (Day 197)
Weight reduction (weight loss) from baseline that is ≥ 10% | Baseline (Week 0) through Week 28 (Day 197)
Weight reduction (weight loss) from baseline that is ≥ 15% | Baseline (Week 0) through Week 28 (Day 197)
Change from baseline in body weight (kg) | Baseline (Week 0) through Week 28 (Day 197)
Change from baseline in body mass index (BMI) | Baseline (Week 0) through Week 28 (Day 197)
Change from baseline in waist circumference | Baseline (Week 0) through Week 28 (Day 197)
Occurrence of treatment emergent adverse events (TEAEs) | Baseline (Week 0) through Week 37 (Day 265)
  Treatment emergent adverse events include adverse events of clinical interest as well as abnormal clinical significant physical exams, laboratory findings, and 12-lead ECG measurements that meet the definition for an AE.
Minimum observed concentration (Cmin) | Baseline (Week 0) through Week 28 (Day 197)
Area under the concentration versus time curve during the dosing interval (AUC(0-τ)) | Baseline (Week 0) through Week 31 (Day 220)
Maximum observed concentration (Cmax) | Baseline (Week 0) through Week 31 (Day 220)
Time to maximum concentration (Tmax) | Baseline (Week 0) through Week 31 (Day 220)
Percent change from baseline in body weight at all protocol-specified post-baseline measurements during the exploratory extension study | Week 28 to Week 60
Occurrence of treatment emergent adverse events (TEAEs) during the exploratory extension study | Week 28 to Week 60
  Week 28 to Week 60

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Research Site MET097 24-201-001, Anaheim, California
  - Research Site MET097 24-201-002, Hollywood, Florida

IPD SHARING:
Plan to Share IPD: Undecided